CLINICAL TRIAL: NCT06138717
Title: The Effect of Aerobic Exercises and Yoga Exercises on Spinal Mobility, Functional Capacity and Disease Activity in Axial Spondyloarthritis: a Randomized Controlled Trial
Brief Title: The Effect of Aerobic Exercises and Yoga Exercises in Axial Spondyloarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Refiye000000000000000000000002
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Axial Spondyloarthritis and Ankylosing Spondylitis
Keywords: Axial spondyloarthritis, yoga, aerobic exercise
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- only aerobic exercise (Active Comparator): Aerobic exercises will be performed with a lower extremity ergometer for 30 minutes and 12 sessions.
  Interventions: Other: yoga based exercises
- combine aerobic exercise and yoga exercises (Active Comparator): Aerobic exercises will be performed with a lower extremity ergometer for 30 minutes and 12 sessions.A yoga-based exercise programme consisting of exercises will be applied for 40 minutes and 12 session
  Interventions: Other: yoga based exercises

INTERVENTIONS:
Other: yoga based exercises — Aerobic exercises will be performed with a lower extremity ergometer for 30 minutes and 12 sessions.In group 2, in addition to aerobic exercises, spinal stretching, relaxation, respiration and meditation will be performed. A yoga-based exercise programme consisting of exercises will be applied for 40 minutes and 12 session
  Other Names: aerobic exercises

SUMMARY:
Axial Spondyloarthritis (AxSpA), mainly affecting the axial skeleton and sacroiliac joints, is a chronic, systemic, inflammatory disease that causes structural and functional disorders. Exercise has a significant role to play in managing treatments. This study aimed to determine the effect of yoga-based exercises combined with aerobic exercise on spinal mobility, disease activity and aerobic capacity in AxSpA.

DETAILED DESCRIPTION:
The study included 60 AxSpA patients according to ASAS criteria. Patients will be divided into two groups randomised. Group 1 (n=30) received only aerobic exercise, group 2 (n=30) received aerobic exercise and yoga exercises will be applied. Aerobic exercise intensity will be measured by cardiopulmonary exercise test (CPET). determined.

Aerobic exercises will be performed with a lower extremity ergometer for 30 minutes and 12 sessions. In group 2, in addition to aerobic exercises, spinal stretching, relaxation, respiration and meditation will be performed. A yoga-based exercise programme consisting of exercises will be applied for 40 minutes and 12 sessions.

Functional capacity before and after treatment, 6-min walk test (6MWT) and VO2 maximum and disease activity will be assessed by ASDAS-CRP. Clinical measurements Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Metrology Index (BASMI), Ankylosing Spondylitis Quality of Life (ASQL) scale will be used. Fibromyalgia symptom severity scale and widespread pain index scores will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Axial spondyloarthritis patients according to ASAS criteria having a stable health condition, having ongoing fatigue, dyspnea, decreased stamina, difficulty in activities of daily living, anxiety, or depression complaints

Exclusion Criteria:

* Hemodynamically unstable, cardiac and pulmonary system unstable, with neurological, and psychological disorders patients

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
VO2 max | six week
  VO2 max is the maximum rate of oxygen consumption attainable during physical exertion
Six minute walk test | six week
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity

SECONDARY OUTCOMES:
BASMI | six week
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) is an index comprising 5 measures of spinal and hip mobility in AS

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No